CLINICAL TRIAL: NCT05270499
Title: Aveir Single-Chamber Leadless Pacemaker Real-World Evidence Post-Approval Study
Brief Title: Aveir VR Real-World Evidence Post-Approval Study
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10418
Record Dates: First submitted 2022-02-28; First posted 2022-03-08 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Pacemaker; Arrythmia; Bradycardia
Keywords: bradycardia; sick sinus rhythm; pacemaker; av block; Vasovagal Syncope
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Atrioventricular Block; Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single Arm: Non randomized
  Interventions: Device: Aveir VR Leadless Pacemaker System

INTERVENTIONS:
Device: Aveir VR Leadless Pacemaker System — This study will utilize real-world data from patients implanted with the Aveir VR Leadless Pacemaker System. No device intervention will be conducted in this study.

SUMMARY:
The purpose of this post-approval study is to evaluate the long-term safety of the single-chamber Aveir VR leadless pacemaker using real-world evidence methods.

DETAILED DESCRIPTION:
This is a non-randomized, multi-center study leveraging real-world evidence methods that merge multiple real-world datasets from Abbott and the Center for Medicare Services to assess Aveir VR leadless pacemaker safety in a large patient population. The results from this study will data to fulfill the Condition of Approval requirements for the Aveir VR device from FDA.

ELIGIBILITY:
Eligibility Criteria:

* Implanted with an Aveir VR leadless pacemaker
* Continuous enrollment in Medicare Part A and Part B for 12 months prior to implant and for 30 days after implant, except in the case of death within the 30-day period
* Ability to link with Medicare fee-for-service data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had an implant of the Aveir VR device, meet inclusion/exclusion criteria, link to Medicare FFS claims, and survive past 30 days will be included in the analysis
Sampling Method: Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2034-02-28 (Estimated); Study Completion 2034-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Free from Acute Aveir VR System-Related Complications | 30 days
  Freedom from complications through 30 days post implant procedure
Number of Subjects Free from Chronic Aveir VR System-Related Complications | 10 Years
  Freedom from Complications from 31 days through 10 years post implant procedure procedure

SECONDARY OUTCOMES:
Number of Subjects Free from Individual Aveir VR Leadless Pacemaker-Related Complications | 10 Years
  Complication rate of the Aveir VR leadless pacemaker for individual acute and chronic complications
Number of Subjects with End of Device Service Events | 10 Years
  Care of subjects at the end of device service. End-of-device service is defined as any event prior to the 10-year follow-up period which results in the leadless pacemaker being explanted or deactivated, another CIED implanted, or death. All instances of the end-of-service will be summarized by event type and time to event.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott
Locations (1):
- Abbott, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No